CLINICAL TRIAL: NCT00737087
Title: A Multi-centred, Non-comparative, Non-randomised, Open, Post Marketing Investigation to Look at the Long-term Clinical Efficacy of the Delta Xtend Reverse Total Shoulder Used in the Treatment of Shoulders With Rotator Cuff Deficiencies.
Brief Title: Long-term Clinical Effectiveness of the Delta Xtend Reverse Total Shoulder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to low follow-up compliance at study sites.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0515
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Cuff Tear Arthropathy; Osteoarthritis With Cuff Deficiency; Rheumatoid Arthritis; Post Traumatic Injury to Shoulder; Revision Surgery of a Failed Anatomic Shoulder Prosthesis
Keywords: total shoulder replacement; rotator cuff; osteoarthritis; rheumatoid arthritis; Delta Extend
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delta Xtend Reverse Total Shoulder (Other): Orthopaedic implant for total shoulder replacement
  Interventions: Device: Delta Xtend Reverse Total Shoulder

INTERVENTIONS:
Device: Delta Xtend Reverse Total Shoulder — Orthopaedic implant for total shoulder replacement

SUMMARY:
This post-marketing study is designed to collect data relating to the use of the Delta Xtend™ Total Shoulder Replacement System in shoulder with rotator cuff deficiencies. This allows for continued monitoring of the performance and safety of the prosthesis in a broader range of clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged less than 85 years inclusive.
* Subjects who have cuff tear arthropathy, osteoarthritis with cuff deficiency, rheumatoid arthritis, post traumatic injury, or a need for revision surgery of a failed anatomic prosthesis in the left or right shoulder, which requires (total) shoulder arthroplasty.
* Subjects with radiographic evidence of sufficient bone stock to seat and support the Delta XtendÔ Reverse Total Shoulder System.
* Subjects who in the opinion of the Clinical Investigator are considered suitable for treatment with the Delta Xtend Reverse Total Shoulder System.
* Patients with a life expectancy of greater than 12 months.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

Exclusion Criteria:

* Male and female subjects aged 86 years or older.
* Subjects with complete deltoid muscle palsy in the target joint as determined by clinical evaluation.
* Subjects with active local or systemic infection or with a history of general or local infections in the target joint over the past 12 months.
* Subjects with severe deformities, or tumours, that would impair fixation or proper positioning of the implant.
* Subjects with no significant muscle, nerve or vascular disease.
* Subjects with a pathology that, in the opinion of the Clinical Investigator, will adversely affect healing.
* Known allergic reactions to implant materials (e.g. bone cement, metal, polyethylene) implant corrosion or implant wear debris.
* Subjects with a known history of poor compliance to medical treatment.
* Subjects who, in the opinion of the Clinical Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical investigation with an investigational product in the last month.
* Subjects who are currently involved in any injury litigation claims.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-11; Primary Completion 2013-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Postoperative functionality through a difference in Constant Score post-treatment, as compared with pre-treatment results. | 2 years

SECONDARY OUTCOMES:
Postoperative functionality at 12weeks, 1, 2, 5 and 10 years through a difference in the Constant score, ASES score, U-Penn score and EQ-5D as compared with pre-treatment scores. | 12weeks, 1, 2, 5 and 10 years
Determine implant survivorship and surgical revision information at 1, 2, 5 and 10 years via Kaplan-Meier survival analysis. | 1, 2, 5 and 10 years

CONTACTS AND LOCATIONS:
Locations (5):
- Universitair Ziekenhuis, Ghent, Belgium
- France (3):
  - Clinique Generale D'Annecy, Annecy
  - CHRU Reims Hôpital Maison Blanche, Reims
  - Polyclinique de l'Atlantique, Saint-Herblain
- Krankenhaus Munchen Bogenhausen, München, Germany